CLINICAL TRIAL: NCT06183125
Title: Reduce Sedentariness and Enhance Physical and Psychological Health of Office Workers With TCM-based Anti-sedentary Intervention: Efficacy and Potential Psychophysiological Mechanisms
Brief Title: Reduce Sedentariness and Enhance Psychological Well-being of Office Workers With TCM-based Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSANG Hector Wing-Hong, Chair Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V2023
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Sedentary Behavior
Keywords: sedentary behavior; office worker; Traditional Chinese Medicine; RCT; psychophysiological mechanism
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial will be conducted among 64 office workers with self-reported sitting time of 5.5 hours or longer per workday. They will be randomly assigned to intervention (TCM-based program) and wait-list control groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the experiment, participants will not be blinded. However, the intervention provider and the evaluator will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TCM-based anti-sedentariness intervention group (Experimental): TCM-based anti-sedentariness intervention
  Interventions: Behavioral: Traditional Chinese Medicine-based program
- Wait-list control group (Other): After the completion of all evaluations, the intervention content will be administered to the experimental group in the same manner.
  Interventions: Behavioral: Traditional Chinese Medicine-based program

INTERVENTIONS:
Behavioral: Traditional Chinese Medicine-based program — Week1-2: one health talk session(60 mins); three workshops (each workshop will last for 60-90mins) to provide hands-on training in Baduanjin, acupressure techniques, mindful stretching, and effective strategies to combat sedentary behavior in the workplace.
  Week 3-4: group practice sessions will take place for one hour every other day throughout the workweek; website support.
  Other Names: TCM-based program

SUMMARY:
The goal of this clinical trial is to test the effects of a TCM-based anti-sedentariness program on workplace sitting time, perceived stress, and cortisol in office workers.The main questions it aims to answer are:

1. Can a Traditional Chinese Medicine (TCM)-based anti-sedentariness program effectively reduce workplace sitting time, perceived stress and cortisol levels among office workers?
2. Whether such anti-sedentary effect works through stress management and enhances when holistic thinking is endorsed.

Participants will engage in a 4 week TCM-based program intervention including 2 weeks of health education and promotion activities (understanding sedentary behaviors, Baduanjin, acupressure, dantian breathing, and mindfulness) and 2 weeks of supported self-practice (daily reminders and tips, regular feedback on sitting time, and individual consultation).

Researchers will compare a group receiving a Traditional Chinese Medicine (TCM)-based intervention with a wait-list control group to determine the effectiveness of the intervention in reducing sitting time and enhancing physical and psychological health.

DETAILED DESCRIPTION:
Introduction:

Sedentary behaviors and their associated physical and mental health risks among adults have received growing concerns among the clinical and research communities. Office workers commonly engage in sedentary behaviors due to their long stationary hours. Evidence has revealed that higher levels of sedentary behaviors were associated with higher perceived stress levels at workplace. However, scarce studies focused on the role of stress management in reducing sedentary behaviors. Traditional Chinese medicine (TCM)-based body works (such as dantian breathing, qigong, and acupressure) are low-cost techniques and found to be primising in addressing stress and sedentary behaviors at workplace. The health benefits of TCM-based bodywork in sedentary office workers may be enhanced when the workers endorse holistic thinking.

The present research aims to test the effects of a TCM-based anti-sedentariness program on workplace sitting time, perceived stress, and cortisol in office workers. Investigators will also explore the psychophysiological mechanism whether such anti-sedentary effect works through stress management and enhances when holistic thinking is endorsed.

Methods:

A systematic review and meta-analysis has been conducted to synthesize the pooled effect of existing anti-sedentariness interventions on office workers' sitting time and compare the effectiveness of different intervention types in reducing sedentary behaviors relative to the control group. The systematic review and meta-analysis set the theoretical foundation of intervention elements for the reduction of sedentary behaviors at workplace and their psychological effects to be applied in the present study.

A randomized controlled trial will be conducted among 92 office workers with self-reported sitting time of 5.5 hours or longer per workday. Participants will be randomly assigned to intervention (TCM-based program) and wait-list control groups. The TCM-based program will last for 4 weeks, with 2 weeks of health education and promotion activities (understanding sedentary behaviors, Baduanjin, acupressure, dantian breathing, and mindfulness) and 2 weeks of supported self-practice (daily reminders and tips, regular feedback on sitting time, website support and individual consultation). Participants' sitting time per workday and perceived stress will be assessed at baseline, post-intervention (4 weeks after baseline), and follow-up (6 weeks after baseline). During the 2-week self-practice, participants in the intervention group will complete a diary of self-practice duration of TCM-based bodywork, perceived stress, and collect saliva samples every two days. Repeated-measures ANOVA will be used to test the group differences in changes in sitting time and perceived stress. Mediating effects of perceived stress and cortisol and moderating effects of holistic thinking will be explored through SPSS marcos.

Significance:

The findings of this study will provide valuable insights into the effectiveness of a TCM-based intervention in reducing sedentary behavior and improving psychological well-being. It is innovative to understand the psychophysiological mechanism of reducing sedentary behavior to explore tailored interventions to enhance the health quality of office workers. Given the easy practice and low cost of the TCM-based body works, the project can put forward a cost-effective intervention that can benefit a large population sustainably.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or above with a full-time and office-based job
2. Reported >5.5 hours of sitting per day at work
3. Native Chinese speaker (Cantonese or Mandarin)
4. Be able to give consent

Exclusion Criteria:

1. Have severe or chronic illness and not suitable for physical exercise
2. Be oversensitive to tactile stimulation
3. Have regular practice of qigong, acupressure, or mindfulness-based activities during the 4 weeks prior to recruitment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
sedentary behavior- total sitting time/workday | Baseline, week 5, week 9
  measured by Actigraph wGT3X-BT
sedentary behavior- sitting time/9-h working time | Baseline, week 5, week 9
  measured by Actigraph wGT3X-BT
Self-report sedentary behaviors | Baseline, week 5, week 9
  measured by International Physical Activity Questionnaire (IPAQ short version) with 8 items. Physical activity levels can be classified as low intensity when the weekly MET (metabolic equivalent of task) value is less than 600, moderate intensity when it ranges from 600 to 3000 MET, and high intensity when it exceeds 3000 MET per week.
psychological stress | Baseline, week 5, week 9
  measured by perceived stress scale(PSS) with 10 items. Each item in the PSS questionnaire is rated on a five-point Likert scale, ranging from 0 (never) to 4 (very often). Participants are asked to indicate the frequency with which they have experienced each event over the past month.The total score on the PSS can range from 0 to 40. Higher scores indicate a higher level of perceived stress.
physiological stress | Baseline, week 5, week 9
  measured by salivary cortisol concentration(measured in ng/mL)

SECONDARY OUTCOMES:
Holistic thinking | Baseline
  measured by Analysis-Holism Scale (AHS), which consists of 24 items. Items are rated on a scale ranging from 1 to 7 (1 = strongly disagree, 7 = strongly agree). The total score on the AHS can range from 24 to 168. Higher scores indicate greater holistic cognitive style, and lower scores indicate greater analytic cognitive style.
Health-related quality of life | Baseline, week 5, week 9
  measured by The Chinese (Hong Kong) SF-36 Health Survey. It consists of 36 questions that cover eight different domains: physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. A higher score indicates better quality of life.
Sleep quality | Baseline, week 5, week 9
  measured by The Pittsburgh Sleep Quality Index, PSQI.The Pittsburgh Sleep Quality Index consists of 19 individual items, with a total score of 21 and a higher score indicating poorer sleep quality.
Psychological distress | Baseline, week 5, week 9
  measured by Depression Anxiety Stress Scale(DASS).The DASS-21 consists of 21 items, with seven items dedicated to each of the three subscales: depression, anxiety, and stress. A higher score indicates more depression, anxiety and stress.
Self efficay | Baseline, week 5, week 9
  measured by The Chinese Self-Efficacy Scale. It consists of 10 items.The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Blood pressures | Baseline, week 5, week 9
  Systolic and diastolic blood pressure will be measured by Omron blood pressure monitor.
Hand grip strength | Baseline, week 5, week 9
  measured by Jamar handheld dynamometer
IL-6 | Baseline, week 5, week 9
  Collect saliva samples to assay IL-6 concentration by using enzyme-linked immunoassay according to the manufacturer's instruction.

CONTACTS AND LOCATIONS:
Overall Officials: Hector Tsang, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No